CLINICAL TRIAL: NCT05939336
Title: The Prebiotic Potential of a Yeast Cell Wall Fraction Containing Mannooligosaccharides and β-glucans.
Brief Title: MOS Prebiotic Potential in Older Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Lallemand Bio-Ingredients (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB202301046
Record Dates: First submitted 2023-07-03; First posted 2023-07-11 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Healthy
Keywords: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mannooligosaccharides (Experimental): Mannooligosaccharides yeast extract
  Interventions: Dietary Supplement: Mannooligosaccharides yeast extract

INTERVENTIONS:
Dietary Supplement: Mannooligosaccharides yeast extract — 15 g per day of mannooligosaccharide yeast extract.

SUMMARY:
Mannooligosaccharides (MOS) derived from baker's yeast may have prebiotic properties such as improving gastrointestinal function. The aims of this study are to determine the effect of MOS on gastrointestinal function and symptoms and fecal microbiota in older adults.

DETAILED DESCRIPTION:
Novel prebiotics with specific microbiome targets and without adverse gastrointestinal symptoms are needed for the exploration of health benefits. This is a 3-week, open-label pilot study designed to evaluate the effect of 15 g per day of yeast-derived mannooligosaccharides on gastrointestinal symptoms, stool frequency, fecal microbiome, and urinary metabolites.

ELIGIBILITY:
Inclusion Criteria:

* Adults 50-99 years of age.
* Able to provide written informed consent in English.
* Willingness to complete all study procedures
* Healthy or diagnoses with Parkinson's or multiple system atrophy

Exclusion Criteria:

* Yeast allergy.
* Self-reported kidney disease.
* Elite athletes or long-distance runners.
* Use of antibiotic drugs (e.g., neomycin, rifaximin) within 1 month of the screening visit.
* Current use of laxatives or antidiarrheal medications.
* Use of other investigational products within 3 months of the screening visit.
* Previously or currently being treated for any intestinal disease or condition, including IBS, Crohn's disease, ulcerative colitis, celiac disease, or gastrointestinal cancer (self-report).
* Previous gastrointestinal surgery (e.g., gastric bypass, fundoplication, bowel resection)
* Current cancer treatment
* Currently pregnant

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Mean daily rating of gastrointestinal symptoms | 14 days
  Change from baseline mean sum of daily mean rating from 0 (no symptom) to 3 (severe symptoms)

CONTACTS AND LOCATIONS:
Locations (1):
- Food Science and Human Nutrition Department, University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moreno ML, Abbeele PVD, Baudot A, Tompkins TA, Taft DH, Yao R, Auger J, Colee J, Dahl WJ. Yeast mannans promote laxation and specifically modulate microbiota composition in older adults: An open-label pilot study. Nutr Res. 2025 Apr;136:15-27. doi: 10.1016/j.nutres.2025.02.004. Epub 2025 Feb 26. PMID 40117931